CLINICAL TRIAL: NCT04341844
Title: Intraoperative Infusion of Methylene Blue for Prevention of Postoperative Delirium and Cognitive Dysfunction in Elderly Patients Undergoing Major Elective Noncardiac and Nonneurosurgical Surgery
Brief Title: Intraoperative Infusion of Methylene Blue for Prevention of Postoperative Delirium and Cognitive Dysfunction in Elderly Patients Undergoing Major Elective Noncardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jun Zhang, Principal Investigator, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KY2019-274
Record Dates: First submitted 2020-03-31; First posted 2020-04-10 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Postoperative Delirium; Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Emergence Delirium; Postoperative Cognitive Complications | interventions — Methylene Blue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylene Blue (Experimental): 2mg/kg MB diluted with normal saline into total 50 ml volume intravenous administration after induction of anesthesia within one hour.
  Interventions: Drug: Methylene Blue
- Control (Placebo Comparator): normal saline in total 50 ml volume intravenous administration after induction of anesthesia within one hour.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylene Blue — 2mg/kg MB diluted with normal saline into total 50 ml volume intravenous administration after induction of anesthesia within one hour.
  Arms: Methylene Blue
Drug: Placebo — normal saline in total 50 ml volume intravenous administration after induction of anesthesia within one hour.
  Arms: Control

SUMMARY:
Postoperative neurocognitive impairments often occur in elderly patients undergoing anesthesia and non-cardiac surgery, including postoperative delirium (POD) and postoperative cognitive dysfunction (POCD). These disorders are often associated with increased mortality and morbidity, prolonged length of hospital stay, functional and cognitive decline with nursing home or long-term care facility placement. Until now highly effective intervention has not been established yet. As a mitochondrial protective agent, the role of methylene blue(MB) in preventing elderly patients from POD/POCD is unknown.Therefore, investigators design this study to validate its prevention against POD/POCD and the aim of this study is to evaluate the efficacy and safety of perioperative administration of MB for POD/POCD prevention.

DETAILED DESCRIPTION:
Postoperative neurocognitive impairments often occur in elderly patients undergoing major surgery, including postoperative delirium(POD) characterized by an acute change in cognition with altered consciousness and impaired attention, and postoperative cognitive dysfunction(POCD) mainly manifested as reduced ability of learning and memory. POD and POCD are major complications that cause disability and distress for millions of patients annually.In 2004, there was an estimated 5-40% incidence in 7.9 million patients over 65 years who had a surgical procedure subsequently experiencing either POD or POCD.The underlying pathophysiology of Postoperative neurocognitive impairments is increasingly understood, implicating a prominent role of neuroinflammation, oxidative stress and mitochondrial dysfunction.Recent experimental evidences reveal that mitochondrial dysfunction is increasingly considered a significant contributor to the development of POD and POCD.

Methylene blue(MB) is a diaminophenothiazine with a long history of clinical use due to its minimal side effect profiles. MB currently is used for treatment of methemoglobinemia, carbon monoxide poisoning, and vasoplegic syndrome as well as for surgical staining. MB could diffuse rapidly into brain and accumulate in the cytoplasm and mitochondria of neurons. In recent years its role as a mitochondrial protective agent has elicited much of its renewed interest, especially, studies have shown that MB has established its neuroprotective effects against ischemic stroke, post-chemotherapy-induced Encephalopathy and neurodegenerative diseases caused by Alzheimer's disease(AD) and psychoses.To date, there is no trials have examined the role of intraoperative MB administration in prevention of POD and POCD in elderly patients undergoing non-cardiac surgery, who have preoperative normal neurocognitive function. Therefore, investigators design this study to evaluate the efficacy and safety of perioperative administration of MB for POD/POCD prevention. It's an entirely novel therapy for postoperative neurocognitive disorders and will have high clinical translatable value if this intervention is found to be beneficial.

ELIGIBILITY:
Inclusion Criteria:

* aged 60-80 years old
* planning to undergo non-cardiac and non-neurosurgical surgery (e.g..thoracic, orthopaedic, urologic and major abdominal surgeries) under general anesthesia
* MMSE>20
* Liver and kidney function are normal
* Patients have the ability to act in full spirit, understand and sign the informed consent, and are willing to complete the whole research process.

Exclusion Criteria:

* Patients with personal history of allergy to methylene blue
* Emergency Surgery
* Patients have 6-phospho-glucose dehydrogenase deficiency (vicia faba disease)
* Patients have recent drug administration that may lead to drug interactions(e.g..SSRIs, SNRIs)
* Patient with a history of major head trauma
* Patients with a history of drug or alcohol abuse
* Patient has serious mental or neurological disorders
* Patients with severe language, hearing and visual impairment
* Patients have serious medical diseases(e.g..heart failure, acute stage of myocardial infarction or respiratory failure)
* Illiteracy
* Patients have participated in other clinical trials in the last 3 months.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative delirium(POD) | Participants will be followed for the duration of hospital stay, an expected average of 5 days.
  the effectiveness of MB in reducing the incidence of POD compared with placebo in elderly patients undergoing major elective non-cardiac surgery.

SECONDARY OUTCOMES:
Incidence of postoperative cognitive dysfunction (POCD) | Up to 3 month after surgery
  the effectiveness of MB in reducing the incidence of POCD compared with placebo in elderly patients undergoing major elective non-cardiac surgery.
Safety Assessments: incidence of perioperative adverse events | the whole perioperative period
  the incidence of perioperative adverse events to reflect safety of intraoperative intravenous 2mg/kg MB administration
Oxidative Stress Biomarkers | the day before surgery and postoperative one day
  the Changes in levels of oxidative stress biomarkers( superoxide dismutase(SOD) and homocysteine(HCY) )

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, PhD, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Deiner S, Luo X, Lin HM, Sessler DI, Saager L, Sieber FE, Lee HB, Sano M; and the Dexlirium Writing Group; Jankowski C, Bergese SD, Candiotti K, Flaherty JH, Arora H, Shander A, Rock P. Intraoperative Infusion of Dexmedetomidine for Prevention of Postoperative Delirium and Cognitive Dysfunction in Elderly Patients Undergoing Major Elective Noncardiac Surgery: A Randomized Clinical Trial. JAMA Surg. 2017 Aug 16;152(8):e171505. doi: 10.1001/jamasurg.2017.1505. Epub 2017 Aug 16. PMID 28593326
- [Result] Avidan MS, Maybrier HR, Abdallah AB, Jacobsohn E, Vlisides PE, Pryor KO, Veselis RA, Grocott HP, Emmert DA, Rogers EM, Downey RJ, Yulico H, Noh GJ, Lee YH, Waszynski CM, Arya VK, Pagel PS, Hudetz JA, Muench MR, Fritz BA, Waberski W, Inouye SK, Mashour GA; PODCAST Research Group. Intraoperative ketamine for prevention of postoperative delirium or pain after major surgery in older adults: an international, multicentre, double-blind, randomised clinical trial. Lancet. 2017 Jul 15;390(10091):267-275. doi: 10.1016/S0140-6736(17)31467-8. Epub 2017 May 30. PMID 28576285
- [Result] Tucker D, Lu Y, Zhang Q. From Mitochondrial Function to Neuroprotection-an Emerging Role for Methylene Blue. Mol Neurobiol. 2018 Jun;55(6):5137-5153. doi: 10.1007/s12035-017-0712-2. Epub 2017 Aug 24. PMID 28840449
- [Result] Gonzalez-Lima F, Barksdale BR, Rojas JC. Mitochondrial respiration as a target for neuroprotection and cognitive enhancement. Biochem Pharmacol. 2014 Apr 15;88(4):584-93. doi: 10.1016/j.bcp.2013.11.010. Epub 2013 Dec 4. PMID 24316434